CLINICAL TRIAL: NCT01015326
Title: Development of a Functional Assessment of Side-effects to Therapy (FAST) Questionnaire to Assess Dermatology-Related Quality of Life in Patients Treated With EGFR Inhibitors: The FAST-EGFR Inhibitors: The FAST-EGFRI and Development of an Investigator Grading System: The Skin and Eye Reactions to Inhibitors of EGFR (SERIES) Score
Brief Title: Development of Dermatology-related Quality of Life Assessment in Patients Treated With Epidermal Growth Factor Receptor (EGFR) Inhibitors
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology and Pediatrics, Northwestern University
Other Study IDs: 1918-004
Record Dates: First submitted 2009-11-06; First posted 2009-11-18 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Skin Toxicities
Keywords: EGFRI; HRQL; Quality of Life; Development of a standardized HRQL instrument for anti-EGFR therapy induced
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Expert Interviews: Expert cohort consists of providers with expertise in administering epidermal growth factor receptor inhibitors (EGFRI) or treating patients with EGFRI-associated skin toxicities. Experts will be asked open-ended questions about symptoms and issues as they relate to HRQL in patients with EFGRI skin toxicities. Experts will then be presented with a pool of potential items and will be asked through interview and questionnaire to relate items according to how common and how important they are when occurring in patients with this condition.
  Interventions: Other: Questionnaire
- Patient Interviews: Patient cohort will consist of those treated with an epidermal growth factor receptor inhibitor (EGFRI) and referred to a specialized dermatology clinic for skin rash management. Patients will be asked open-ended questions about symptoms and issues as they relate to their HRQL to elicit personal experiences about how EGFRI skin toxicities and its treatment affects patients. Patients will be asked through interview and questionnaire to rate items according to how often they are experienced and how important they are to the patient.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Administered questionnaire
  Groups: Expert Interviews
Other: Questionnaire — Administered questionnaire
  Groups: Patient Interviews

SUMMARY:
Epidermal Growth Factor Receptor Inhibitors (EGFRI) are associated with skin toxicities. Clinical experience suggests that skin toxicities interfere with health related quality of life (HRQL) and may interfere with treatment adherence. No systematic investigations of EGFRI-associated dermatologic toxicities and impact on HRQL have been reported. No patient-reported outcome measures exist to capture the unique concerns of oncology patients who experience EGFRI-associated dermatologic toxicities.

The purpose of this study is to develop a patient-reported outcomes measure to assess dermatologic-related symptoms burden and health-related quality of life among patients receiving an EGFRI, and to develop a grading system for EGFRI-associated dermatologic toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing anti-EGFR cancer therapy
* Over 18 years old

Exclusion Criteria:

* Unable to complete the questionnaire
* Unable to follow instructions or give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an EGFRI and referred to a specialized dermatology clinic for skin rash management.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P West, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Expert Interviews: Expert cohort consists of providers with expertise in administering epidermal growth factor receptor inhibitors (EGFRI) or treating patients with EGFRI-associated skin toxicities. Experts will then be presented with a pool of potential items and will be asked through interview and questionnaire to relate items according to how common and how important they are when occurring in patients with this condition.
  Questionnaire : Administered questionnaire
- Patient Interviews: Patient cohort will consist of those treated with an epidermal growth factor receptor inhibitor (EGFRI) and referred to a specialized dermatology clinic for skin rash management. Patients will be asked through interview and questionnaire to rate items according to how important they are to the patient's health-related quality of life (HRQL).
  Questionnaire : Administered questionnaire
Period: Overall Study
Arm/Group | Expert Interviews | Patient Interviews
Started | 12 | 20
Completed | 11 | 18
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Expert Interviews: Expert cohort consists of providers with expertise in administering epidermal growth factor receptor inhibitors (EGFRI) or treating patients with EGFRI-associated skin toxicities. Experts will be asked open-ended questions about symptoms and issues as they relate to health-related quality of life (HRQL) in patients with EFGRI skin toxicities. Experts will then be presented with a pool of potential items and will be asked through interview and questionnaire to relate items according to how common and how important they are when occurring in patients with this condition.
  Questionnaire : Administered questionnaire
- Patient Interviews: Patient cohort will consist of those treated with an epidermal growth factor receptor inhibitor (EGFRI) and referred to a specialized dermatology clinic for skin rash management. Patients will be asked open-ended questions about symptoms and issues as they relate to their health-related quality of life (HRQL) to elicit personal experiences about how EGFRI skin toxicities and its treatment affects patients. Patients will be asked through interview and questionnaire to rate items according to how often they are experienced and how important they are to the patient.
  Questionnaire : Administered questionnaire
- Total: Total of all reporting groups
Arm/Group | Expert Interviews | Patient Interviews | Total
Number analyzed (Participants) | 12 | 20 | 32
Age, Continuous [Mean (Full Range); unit: years] | 39.2 [25 to 52] | 57.0 [34 to 76] | 50.3 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 22
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Data From Patients and Experts to Measure Anti-EGFR Therapy-specific Health-related Quality of Life (HRQL)
Description: Patients were asked "How important is this symptoms or concern to your quality of life?" They were given a series of items (listed in the table) and instructed to assign each item a numerical value of 0 to 3, where 0 is equivalent to "not at all important" and 3 is equivalent to "extremely important." Experts were asked "How important is this symptom or concern to patients' quality of life?" They were given the same series of items and instructed to assign each item a numerical value of 0 to 3, where 0 is equivalent to "not at all important" and 3 is equivalent to "extremely important." For each item, a mean score was calculated using the values assigned to that item from all patients, and a second mean score was calculated using the values assigned to that item from all experts. An item's mean score may range from 0 to 3, where 0 is equivalent to "not at all important to quality of life" and where 3 is equivalent to "extremely important to quality of life."
Time Frame: at time of questionnaire
Population: Additional items that were variably collected and recorded have been omitted from the data set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Expert Interviews | Patient Interviews
Number analyzed (Participants) | 11 | 18
units on a scale
  My skin condition burns or stings | 2.70 (0.48) | 2.41 (0.94)
  My skin hurts | 2.70 (0.48) | 2.29 (1.18)
  My eyes are dry | 1.90 (0.14) | 2.14 (1.17)
  My skin condition affects how well I sleep | 2.40 (0.84) | 2.13 (1.13)
  My skin is flaky and dry | 1.70 (0.67) | 2.00 (1.15)
  My skin itches | 2.20 (0.63) | 2.00 (1.17)
  My skin condition makes it work/hobbies hard | 2.20 (0.79) | 2.00 (1.10)
  My fingers/toes hurt | 2.40 (0.70) | 2.00 (1.07)
  I am satisfied with the condition of my skin | 1.60 (1.17) | 1.94 (0.85)
  I am bothered by increased facial/eyelash hair | 1.70 (0.67) | 1.93 (1.22)
  My skin condition makes me feel depressed | 2.60 (0.70) | 1.88 (1.11)
  My skin condition affects my social life | 2.80 (0.42) | 1.88 (1.09)
  My skin condition bothers me | 1.80 (1.03) | 1.88 (0.89)
  My skin condition makes daily life difficult | 2.00 (0.67) | 1.80 (1.08)
  I am frustrated by my skin condition | 1.60 (0.84) | 1.75 (1.13)
  My skin condition affects my mood | 1.80 (0.92) | 1.71 (1.18)
  I tend to do things by myself because of my skin | 1.90 (0.99) | 1.71 (1.14)
  I tend to stay at home because of my skin | 2.60 (0.52) | 1.60 (1.30)
  I experience pain in certain body parts | 1.90 (0.74) | 1.50 (0.97)
  My skin makes showing affection difficult | 1.90 (1.10) | 1.46 (1.20)
  My skin is a problem for the people I love | 2.00 (0.82) | 1.68 (1.31)

ADVERSE EVENTS:
Arm/Group | Expert Interviews | Patient Interviews
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/20
Other Adverse Events (participants affected / at risk) | 0/12 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes